CLINICAL TRIAL: NCT00818740
Title: Pharmacokinetics of ORM-12741 After Intravenous and Oral Administration and Effects of Food on ORM-12741 Pharmacokinetics; An Open, Randomised, Single Dose, Single Centre, Crossover Study in Healthy Male Subjects
Brief Title: Pharmacokinetic Study of ORM-12741 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Mononen/Clinical Study Manager, R&D
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 3098003
Record Dates: First submitted 2008-12-22; First posted 2009-01-08 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — ORM-12741

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ORM-12741 i.v. (Experimental)
  Interventions: Drug: ORM-12741
- ORM-12741 oral solution (Experimental)
  Interventions: Drug: ORM-12741
- ORM-12741 oral capsule with food (Experimental)
  Interventions: Drug: ORM-12741
- ORM-12741 oral capsule without food (Experimental)
  Interventions: Drug: ORM-12741

INTERVENTIONS:
Drug: ORM-12741 — i.v., oral solution and oral capsule forms. Oral capsule given with and without food.

SUMMARY:
The purpose of this study is to determine pharmacokinetic parameters of ORM-12741 in healthy volunteers.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent (IC) obtained.
* Good general health ascertained by detailed medical history and physical examinations.
* Finnish speaking males between 18 and 45 years of age (inclusive).
* Body Mass Index (BMI) between 18-30 kg/m2 (inclusive, BMI = weight/height2).
* Weight of 55-100 kg (inclusive).

Exclusion criteria:

* A predictable poor compliance or inability to communicate well with the investigator.
* Veins unsuitable for repeated venipuncture.
* Evidence of clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric disease as judged by the investigator.
* Any condition requiring regular concomitant medication including herbal products or likely to need any concomitant treatment during the study.
* Susceptibility to severe allergic reactions.
* Intake of any medication that could affect the outcome of the study, within 2 weeks prior to the first study treatment administration or less than 5 times a half-live of the medication. Possible enzyme inducing drugs will be discussed case-by-case with the sponsor.
* Regular consumption of more than 21 units of alcohol per week (1 unit = 4 cl spirits, about 13 g of alcohol).
* Current use of nicotine-containing products more than 5 cigarettes or equivalent/day.
* Inability to refrain from using nicotine-containing products during the stay at the study centre.
* Inability to refrain from consuming caffeine-containing beverages during the stay at the study centre e.g. propensity in getting headache when refraining from caffeine-containing beverages.
* Blood donation or loss of significant amount of blood within 2 months prior to the screening visit.
* Abnormal 12-lead ECG finding of clinical relevance after 10-minute rest in supine position at the screening visit, for example:
* QTc (calculated through the Bazett's formula) > 450msec,
* PR < 120 msec or > 210 msec,
* QRS < 70 msec or > 120 msec.
* HR < 45 beats/minute or > 100 beats/minute after 10-minute rest in supine position at the screening visit.
* At the screening visit systolic blood pressure (BP) < 90 mmHg or > 140 mmHg after 10 minutes in supine position, diastolic BP < 50 mmHg or > 90 mmHg after 10 minutes in supine position.
* Any abnormal value of laboratory, vital signs, physical examination, which may in the opinion of the investigator interfere with the interpretation of the test results or cause a health risk for the subject if he takes part into the study.
* History of drug abuse or positive result in drug abuse test.
* Positive serology to human immunodeficiency virus antibodies (HIVAgAb), hepatitis C virus antibodies (HCVAb) or hepatitis B surface antigen (HBsAg).
* Any other condition that in the opinion of the investigator would interfere with the evaluation of the results or constitute a health risk for the study subject.
* Participation in a clinical drug study within 3 months prior to the first study treatment administration of this study or earlier participation in a clinical study with ORM-12741.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables including: Peak concentration in plasma (Cmax), Time to peak concentration in plasma (tmax), Area under the plasma concentration-time curve (AUC) | 96 hours

SECONDARY OUTCOMES:
Safety variables including blood pressure (BP), heart rate (HR), electrocardiograms (ECGs), physical examination, laboratory safety variables (haematology, chemistry, serology and urinalysis) and adverse events (AEs). | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Juha Peltonen, MD, Principal Investigator — CRST; Virpi Mononen, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- CRST, Turku, Finland